CLINICAL TRIAL: NCT00866489
Title: Clinical Trial Cencer, Xijing Hospital, Fourth Military Medical University
Brief Title: The Neuroprotective Effects of RPC on the Neurosurgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Hailong Dong, Xijing Hospital, Fourth Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DONG2008RPC
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2009-03

CONDITIONS: s100b
Keywords: Experimental

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sham RIPC (No Intervention): Patients had a deflated cuff placed on the right upper arm for 30 min.
- RIPC (Experimental): RIPC consisted of three 5-min cycles of right upper arm ischemia, which was induced by an automated cuff-inflator placed on the right upper arm and inflated to 200 mmHg, with an intervening 5 min of reperfusion during which the cuff was deflated
  Interventions: Procedure: remote preconditioning

INTERVENTIONS:
Procedure: remote preconditioning — Remote ischemic preconditioning consist of three 5-min cycles of right upper limb ischaemia, induced by an automated cuff-inflator placed on the upper arm and inflated to 200 mm Hg, with an intervening 5 min of reperfusion during which the cuff is deflated.
  Other Names: remote ischemic preconditioning; RIPC
  Arms: RIPC

SUMMARY:
The current study is designed to clarify the neuroprotective effect of remote ischemic precondtioning on the patients underwent neurosurgery.

DETAILED DESCRIPTION:
BACKGROUND: Brain ischemia and injury are commonly contributed to perioperative morbidity and mortality after neurosurgery. Remote ischemic preconditioning (RIPC) is a phenomenon whereby brief periods of ischemia followed by reperfusion in one organ provide systemic protection from prolonged ischemia. To investigate whether remote preconditioning protects the brain injury in patients undergoing elective neurosurgery, a randomized trial will be performed in current study.

DESIGNING Thirty patients undergoing craniotomy for supratentorial meningioma will be randomize assigned to neurosurgery with RIPC or conventional neurosurgery (control). Remote ischemic preconditioning consist of three 5-min cycles of right upper limb ischaemia, induced by an automated cuff-inflator placed on the upper arm and inflated to 200 mm Hg, with an intervening 5 min of reperfusion during which the cuff is deflated. Cerebral injury was assessed by S-100b, NSE, and neurological function scores in different time points.

EXPECTED RESULTS RIPC will reduce the incidence of cerebral injury.

CONCLUSIONS:

In patients undergoing elective craniotomy for supratentorial meningioma, RIPC reduces the incidence of postoperative cerebral injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for primary elective neurosurgery were invited to participate in the study at the time of scheduling for operation

Exclusion Criteria:

* Potential participants were excluded if they were >70 years of age
* Required concomitant procedures other than neurosurgery
* Had experienced an acute coronary syndrome or myocardial infraction within 3 months
* Were unable to give informed consent
* Were taking sulfonylurea oral hypoglycemic agents or nicorandil drug therapy because these agents have been shown to effect preconditioning.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
S-100b and NSE level | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Hailong DONG, M.D.,Ph.D., Principal Investigator — Xijing Hospital